CLINICAL TRIAL: NCT04571242
Title: Open-Label, Post Market Study: Study the Effects of Differential Target Multiplexed Spinal Cord Stimulation (DTM™SCS) Programs in Treating Intractable Chronic Back Pain in Subjects Without Prior History of Spine Surgery
Brief Title: SCS Programming Study in Treating Intractable Chronic Back Pain (NOVA)
Acronym: NOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SGX Nova LLC (Industry)
Responsible Party: Sponsor
Organization: SGX Medical LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTM-NOVA-2020PM1
Record Dates: First submitted 2020-09-02; First posted 2020-09-30 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Chronic Back Pain

STUDY DESIGN:
Intervention Model Description: Subjects meeting study entrance criteria will be randomized in a 1:1 ratio to one of two study treatment groups:
  * Test treatment group with DTM-SCS programming approach
  * Control treatment group with Conventional SCS programming approach
  Data at follow-up visits will be compared between the two treatment groups, and in reference to baseline assessments collected at the beginning of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- DTM-SCS programming (Active Comparator): This SCS group will be programmed under the direction of physicians with support of clinical representatives of the Test treatments, which may identify the type of treatment to study participants. DTM-SCS programming has at least two programs with different pulse rate in the 50 to 1,000 Hz range and each having a maximum pulse width of 1 ms.
  Interventions: Device: DTM Programming
- Conventional SCS programming (Active Comparator): This SCS group will be programmed under the direction of physicians with support of clinical representatives of the Control treatments, which may identify the type of treatment to study participants. Conventional SCS programming is stimulation parameters in the 40-250 Hz frequency range and will be trialed according to standard practice as described in the Intellis labeling/manuals
  Interventions: Device: Conventional SCS programming

INTERVENTIONS:
Device: DTM Programming — DTM-SCS programming
  Arms: DTM-SCS programming
Device: Conventional SCS programming — Conventional SCS programming
  Arms: Conventional SCS programming

SUMMARY:
This is an open-label prospective, randomized, controlled, multi-center study comparing DTM-SCS programming approach to Conventional SCS programming approach.

The purpose of this investigational study is to study the effects of Differential Target Multiplexed Spinal Cord Stimulation (DTM-SCS) in subjects with chronic, intractable pain of the trunk with or without lower limb pain, including unilateral or bilateral pain without prior history of spine surgery and refractory to conservative and surgical interventions.

DETAILED DESCRIPTION:
This is an open-label prospective, randomized, controlled, multi-center study comparing DTM-SCS programming approach to Conventional SCS programming approach.

Subjects meeting study entrance criteria will be randomized in a 1:1 ratio to one of two study treatment groups:

* Test treatment group with DTM-SCS programming approach
* Control treatment group with Conventional SCS programming approach

Data at follow-up visits will be compared between the two treatment groups, and in reference to baseline assessments collected at the beginning of the study.

There is an optional two-way crossover to the other treatment group available for all subjects who remain implanted at 6 month visit.

Up to 250 subjects may be enrolled at up to 20 clinical sites in the United States in order to include an estimated 135 subjects to the point of randomization.

This would allow a minimum of 100 subjects (50% in each treatment arm) to complete the 3-month endpoint.

The expected total duration of this study is approximately 32 months.

ELIGIBILITY:
Inclusion Criteria:

1. Be a candidate for SCS system (trial and implant) per labeled indication (back pain with or without leg pain)
2. Have been diagnosed with chronic, refractory axial low back pain with a neuropathic component and are not eligible for spine surgery (e.g., lumbar fusion, discectomy, laminectomy, laminotomy) at the time of enrollment
3. Has an average back pain intensity ≥ 6.0 cm on the 10.0 cm Visual Analog Scale (VAS) at the time of enrollment
4. Be willing and capable of giving written informed consent to participate in this clinical study based on voluntary agreement after a thorough explanation of the subject's participation has been provided.
5. Be willing and capable of subjective evaluation, read and understand written questionnaires, and read, understand and sign the written inform consent.
6. Be 18 years of age or older at the time of enrollment
7. Be on a stable pain medication regimen, as determined by the study investigator, for at least 30 days prior to enrolling in this study
8. Be willing to not increase pain medications from baseline through the 3-Month Visit
9. Be willing and able to comply with study-related requirements, procedures, and visits

Exclusion Criteria:

1. Had previous lumbar spinal surgery (e.g., lumbar fusion, discectomy, laminectomy, laminotomy)
2. Has a medical, anatomical, and/or psycho-social condition that is contraindicated for commercially available Intellis™ SCS systems as determined by the Investigator
3. Has a diagnosed back condition with inflammatory causes of back pain (e.g., onset of severe pain with activity), serious spinal pathology and or neurological disorders, as determined by the Investigator
4. Be concurrently participating in another clinical study
5. Has an existing active implanted device such as a pacemaker, another SCS unit, peripheral nerve stimulator and/or drug delivery pump, etc.
6. Has a pain in other area(s) and/or medical condition requiring the regular use of significant pain medications that could interfere with accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the Investigator
7. Has mechanical spine instability as determined by the Investigator
8. Has undergone, within 30 days prior to enrollment, an interventional procedure and/or surgery to treat back and/or leg pain, which is providing significant pain relief
9. Has unresolved major issues of secondary gain (e.g., social, financial, legal), as determined by the investigator
10. Be involved in an injury claim under current litigation or has a pending or approved worker's compensation claim
11. Be pregnant (determined by urine testing unless female subject is surgically sterile or post-menopausal. If female, sexually active, and childbearing age, subject must be willing to use a reliable form of birth control.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Vallejo, MD, Study Chair — SGX Medical
Locations (1):
- SGX Medical, Bloomington, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 121 subjects met inclusion and exclusion criteria after enrollment were randomized (5 subjects failed screening). 105 subjects successfully randomized subjects completed the trial phase and were included in the Modified Intent to Treat Analysis.
Groups:
- DTM-SCS Programming Group: DTM-SCS program group has at least two programs with different pulse rate in the 50 to 1,000 Hz range and each having a maximum pulse width of 1 ms.
- Conventional SCS Programming Group: Conventional SCS program group has stimulation parameters in the 40-250 Hz frequency range will be trialed according to standard practice as described in the Intellis labeling/manuals.
Period: 3 Months
Arm/Group | DTM-SCS Programming Group | Conventional SCS Programming Group
Started | 51 | 54
Completed | 46 | 44
Not Completed | 5 | 10
Period: 6 Months
Arm/Group | DTM-SCS Programming Group | Conventional SCS Programming Group
Started | 46 | 44
Completed | 42 | 43
Not Completed | 4 | 1
Period: 9 Months
Arm/Group | DTM-SCS Programming Group | Conventional SCS Programming Group
Started | 56 (14 subjects from Conventional-SCS crossed over to DTM-SCS after the 6 months visit.) | 29 (0 subjects from DTM-SCS programming crossed over to Conventional SCS programming.)
Completed | 56 | 28
Not Completed | 0 | 1
Period: 12 Months
Arm/Group | DTM-SCS Programming Group | Conventional SCS Programming Group
Started | 56 | 28
Completed | 55 | 28
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTM-SCS Programming Group | Conventional SCS Programming Group | Total
Number analyzed (Participants) | 51 | 54 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (13.5) | 59.6 (12.1) | 61.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 22 | 21 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 51 | 54 | 105
Back Pain VAS [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Score (0.0cm to 10.0cm). Higher score represents more pain.
  units on a scale | 7.9 (1.0) | 8.0 (1.1) | 8.0 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Respond to DTM-SCS Therapy Compared to Conventional SCS Therapy
Description: The primary outcome measure is the percentage of randomized subjects (who completed the trial phase) who respond to SCS therapy at 3-months after device activation. An individual responder is a subject that experiences at least a 50% decrease in back pain relative to baseline assessment.
Time Frame: 3 months
Population: Modified Intent to Treat (mITT): All successfully randomized subjects who complete the Trial Phase. Failed trial subjects and subjects that withdrew due to insufficient pain relief carry forward.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DTM-SCS Programming Group | Conventional SCS Programming Group
Number analyzed (Participants) | 46 | 44
percentage of participants | 93.5 [81.6 to 97.9] | 36.4 [23.6 to 51.4]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- DTM-SCS Programming Group: DTM-SCS program group has at least two programs with different pulse rate in the 50 to 1,000 Hz range and each having a maximum pulse width of 1 ms. All reported adverse events occurred prior to the optional crossover.
- Conventional SCS Programming Group: Conventional SCS program group has stimulation parameters in the 40-250 Hz frequency range will be trialed according to standard practice as described in the Intellis labeling/manuals. All reported adverse events occurred prior to the optional crossover.
Arm/Group | DTM-SCS Programming Group | Conventional SCS Programming Group
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/54
Serious Adverse Events (participants affected / at risk) | 1/51 | 2/54
Other Adverse Events (participants affected / at risk) | 0/51 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTM-SCS Programming Group (N=51) | Conventional SCS Programming Group (N=54)
Spinal Epidural Hematoma (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Post Dural Puncture Headache (Nervous system disorders) | 0 (0) | 1 (1)
Pocket Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT04571242/Prot_SAP_000.pdf